CLINICAL TRIAL: NCT02632357
Title: Longitudinal Experimental Study on ULNTT1 and Cervico-Thoracic Spine Motion Patterns Relationship
Brief Title: Longitudinal Experimental Study on ULNTT and Cervico-Thoracic Spine Motion Patterns Relationship
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Massimo Rossi, MD, University of Milano Bicocca
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UMilanoBicocca
Record Dates: First submitted 2015-12-03; First posted 2015-12-16 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Cervicobrachial Neuralgia
Keywords: Neurodynamics
MeSH Terms: conditions — Brachial Plexus Neuritis | interventions — Manipulation, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AS group (Experimental): Subjects with ULNTT asymmetry > 10°
  Interventions: Other: Spinal Manipulation
- S group (No Intervention): Subjects with ULNTT symmetry

INTERVENTIONS:
Other: Spinal Manipulation
  Arms: AS group

SUMMARY:
Study Design: Longitudinal Experimental Study

Objective: Analyze the relationship between Upper Limb Neural Tension Test (ULNTT1) and cervico-thoracic spine biomechanics using a new motion-capture spine movement data analyzing model based on Least Square Approximation.

Summary of Background Data: ULNTT1 is a test able to determine cervical nerve roots and brachial plexus displacement within their interface structures. No studies were conducted about ULNTT1 and cervico-thoracic spine motion patterns relationship.

Methods: 12 subjects with ULNTT1 asymmetry > 10° (AS group) and 11 subjects with ULNTT1 symmetry (S group) at clinical tests will be enrolled for the study. Subjects will be analyzed for ULNTT1 with an electrogoniometer using two parameters, one operator and one patient-dependent. Fine lateral bending cervico-thoracic spine motion patterns will be collected with motion-capturing technique and data will be analyzed with Least Square Approximation tools. Subjects with impairments in cervico-thoracic spine mobility will undergo to correction of those with spinal manipulative therapy. ULNTT1 and spine mobility will be so re-evaluated with same methods.

ELIGIBILITY:
Inclusion Criteria:

* AS group: ULNTT asymmetry >10°
* S group: ULNTT symmetry

Exclusion Criteria:

* History of neck, shoulder or arm surgical interventions or major trauma, peripheral neuropathy, mental disturbance, limitation of shoulder, elbow or wrist range of motion, BMI >25.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Upper Limb Neural Tension Test at baseline: R2 | Baseline
  ULNTT are neurodynamics test of brachial plexus. Two parameters are collected during the procedure: firm resistance to elbow extension, named R2, operator dependent, and severe pain onset, named P2, patient dependent. Both results are expressed as degrees that left to full elbow extension. Four repetition per side are performed and average value is calculated.
Upper Limb Neural Tension Test at baseline: P2 | Baseline
  ULNTT are neurodynamics test of brachial plexus. Two parameters are collected during the procedure: firm resistance to elbow extension, named R2, operator dependent, and severe pain onset, named P2, patient dependent. Both results are expressed as degrees that left to full elbow extension. Four repetition per side are performed and average value is calculated.
Cervico-Thoracic Spine Lateral Bending at baseline | Baseline
  Cervico-thoracic spine side bending is registered with motion-capture technology. Results are analyzed with Least Square Approximation tools and expressed as mathematical parameters in angles. Four repetition per side are performed and average value is calculated.
Upper Limb Neural Tension Test after intervention: R2 | Immediately after intervention, same day than baseline acquisition
  ULNTT are neurodynamics test of brachial plexus. Two parameters are collected during the procedure: firm resistance to elbow extension, named R2, operator dependent, and severe pain onset, named P2, patient dependent. Both results are expressed as degrees that left to full elbow extension. Four repetition per side are performed and average value is calculated.
Upper Limb Neural Tension Test after intervention: P2 | Immediately after intervention, same day than baseline acquisition
  ULNTT are neurodynamics test of brachial plexus. Two parameters are collected during the procedure: firm resistance to elbow extension, named R2, operator dependent, and severe pain onset, named P2, patient dependent. Both results are expressed as degrees that left to full elbow extension. Four repetition per side are performed and average value is calculated.
Cervico-Thoracic Spine Lateral Bending after intervention | Immediately after intervention, same day than baseline acquisition
  Cervico-thoracic spine side bending is registered with motion-capture technology. Results are analyzed with Least Square Approximation tools and expressed as mathematical parameters in angles. Four repetition per side are performed and average value is calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Zucchi, Carate Brianza, MB, Italy

IPD SHARING:
Plan to Share IPD: No